CLINICAL TRIAL: NCT06531928
Title: The Effect of Chest Tube Withdrawal on Patients' Anxiety Levels After Video-Assisted Thoracoscopic Surgery
Brief Title: Effect of Chest Tube Withdrawal on Patients' Anxiety Levels After Thoracic Surgery
Status: Recruiting | Type: Observational
Sponsor: Ankara Ataturk Sanatorium Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Ramazan Baldemir, Associate Proffessor, Ankara Ataturk Sanatorium Training and Research Hospital
Other Study IDs: 2024-BCEK/61
Record Dates: First submitted 2024-05-28; First posted 2024-08-01 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2025-01

CONDITIONS: Chest Tube Withdrawal; Video-assisted Thoracoscopic Surgery
Keywords: Chest tube withdrawal; Pain; Anxiety; Video-assisted thoracoscopic surgery; VATS
MeSH Terms: conditions — Pain; Anxiety Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: chest tube withdrawal — The Effect of Chest Tube Withdrawal on Patients' Anxiety Levels in Thoracic Surgery Cases Performed with Video-Assisted Thoracoscopic Surgery

SUMMARY:
Since the removal of the chest tube is a painful procedure, it can cause serious anxiety in patients. Patients state that chest tube removal is among the bad memories they experience. The source of the anxiety may be related to fear and anxiety about the pain caused by the upcoming chest tube removal procedure, or it may be the words they have heard from other patients who have had this experience before. There are a limited number of studies in the literature on anxiety that may occur in patients due to chest tube withdrawal. In addition, studies in the literature did not focus on whether there was a difference between pre-procedure and post-procedure anxiety levels. In this study, it was aimed to investigate the anxiety levels before and after the procedure and the pain levels felt in the patients due to the procedure due to chest tube withdrawal in patients who underwent VATS. In addition, it aimed to investigate whether there is any correlation between pre-procedure anxiety and pain experienced during the procedure. If a correlation is detected, the importance of pre-procedural anxiety management will be better understood, the necessity of interventions such as psychological and pharmacological treatment for anxiety will come to the fore, and new research on this subject will be needed.

ELIGIBILITY:
Inclusion Criteria:

* The ages of 18-65
* BMI between 18-35 kg/m2
* Who have undergone VATS
* Who have a single chest tube inserted during surgery
* who have undergone resection with VATS (wedge resection, segmentectomy, lobectomy)

Exclusion Criteria:

* Who have undergone surgery under emergency conditions,
* Who have undergone thoracotomy, decortication, pleural biopsy,
* Who constantly use anti-inflammatory or analgesic drugs,
* Patients with preoperative chronic pain,
* Who have undergone thoracic surgery before,
* Patients with a history of chest tube insertion and for any reason after surgery (prolonged air leakage),
* Patients whose chest tube has not been removed for more than 7 days,
* Who have undergone pleurodesis
* Patients with psychiatric diagnoses or who use psychiatric drugs
* Who are illiterate will be excluded from the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients between the ages of 18-65, those with a BMI between 18-35 kg/m2, patients who have undergone VATS, patients who have a single chest tube inserted during surgery, patients who have undergone resection with VATS (wedge resection, segmentectomy, lobectomy) will be included in the study.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-08-15 (Actual); Primary Completion 2025-06-15 (Estimated); Study Completion 2025-07-30 (Estimated)

PRIMARY OUTCOMES:
visual analog scale -Anxiety | 24 hours
  Investigation of pre-procedure and post-procedure anxiety levels due to chest tube removal in patients undergoing VATS and pain felt by patients due to the procedure. The VAS-anxiety is a segmented numerical version of the visual analog scale (VAS), in which the respondent chooses an integer (0-100 mm) that best reflects the intensity of his anxiety. It is considered a one-dimensional measure of anxiety intensity in adults. It ranges from "0 mm" representing no anxiety to "100 mm" representing extreme anxiety.

SECONDARY OUTCOMES:
visual analog scale-Pain | 24 hours
  It was aimed to investigate whether there is any correlation between pre-procedure anxiety and pain experienced during the procedure. The VAS-pain is a segmented numerical version of the visual analog scale (VAS), in which the respondent chooses an integer (0-100 mm) that best reflects the intensity of his pain. It is considered a one-dimensional measure of pain intensity in adults. It ranges from "0 mm" representing no pain to "100 mm" representing extreme pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Atatürk Sanatorium Training and Research Hospital, Ankara, Keçiören, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No